CLINICAL TRIAL: NCT03399838
Title: The PedINDex Study: Comparing Intranasal Dexmedetomidine With Oral or Rectal Midazolam for Procedural Sedation in the Pediatric Emergency Department.
Brief Title: Comparing in Dexmedetomidine With po/pr Midazolam for Procedural Sedation in the Pediatric Emergency Department
Acronym: PedINDEX
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor left the hospital
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PedINDEX study
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Procedural Anxiety; Emergencies
Keywords: Procedural Sedation and Analgesia; Pediatric Emergency Department; intranasal; dexmedetomidine; midazolam; anxiety relief
MeSH Terms: conditions — Emergencies; Agnosia | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Intervention Model Description: randomised trial comparing 2 drugs (midazolam, dexmedetomidine)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Application of single dose of 4mcg/kg dexmedetomidine intranasally for pediatric procedural sedation at the emergency department
  Interventions: Drug: Dexmedetomidine
- Midazolam (Active Comparator): 0.5mg po/pr midazolam for pediatric sedation at the emergency department
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — IN Dex for pediatric procedural sedation at the emergency department
  Arms: Dexmedetomidine
Drug: Midazolam — po/pr midazolam as active comparator to dexmedetomidine for pediatric procedural sedation at the pediatric emergency department
  Arms: Midazolam

SUMMARY:
This study aims to compare efficacy of Procedural Sedation with Dexmedetomidine as compared to Midazolam in the pediatric Emergency Department.

210 children aged 6 months to 6 years will be included and randomly assigned to receiving oral or rectal midazolam (standard of care) or intranasal dexmedetomidine for procedures at the emergency department where mainly a sedation and no analgesia is sought. The procedure will be videotaped and analysis is blinded to the medication.

DETAILED DESCRIPTION:
Pediatric sedation and analgesia is a major aspect in emergency procedures and treatments: anxiety and stress in children need to be purposefully addressed in order to perform procedures where a child needs to lie still, and to prevent anxiety in the future. An important factor to reduce stress and anxiety is the use of medication without the need of an intravenous access. To date, options for such a sedation are very limited. One of the most common medications in use is midazolam applied orally or rectally, though there are several concerns with this drug.

Pediatric developmental stage often does not allow to rationally explain procedures (e.g., wound management, emergency radiologic imaging, lumbar punctures, posing a difficult iv line), thus provoking further anxiety and non-compliance.

The medication in question (dexmedetomidine, DEX) has been proven to be a safe and reliable sedative in different settings even though its use is off-label in pediatrics. Data on its use in the pediatric emergency department (PED) are sparse, but it could be of help in a variety of situations especially in this setting.

The overall objective of this study is to determine whether intranasal (IN) DEX has better efficacy profile for PSA in the PED compared to rectal (PR)/ oral (PO) midazolam in children aged 6 months to 6 years.

Validated scores are used to describe efficacy in detail, including Procedural Sedation State Scale, Modified Yale Preoperative Anxiety Scale Short Form, University of Michigan Sedation State. Surveys to the parents and the health care professionals are used to further describe efficacy.

Procedural Sedation State Scale will be the primary outcome. Based on clinical experience we expect around 70% of patients with midazolam sedation to score 2 or 3 using the PSSS (target sedation state). Clinically relevant superiority is defined as 15% more patients with target sedation state.

Study design: single-center, prospective, randomised, active control, rater-blinded trial: procedures will be videotaped and analysed by research assistants blinded to the study medication.

Number of patients: 210 with assessable primary outcome. Duration of recruitment is expected to be 24 months

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 months and 6 years presenting at the pediatric emergency department
* Indication for midazolam as sedation
* Signed informed consent

Exclusion Criteria:

* Contraindication for midazolam
* Contraindication for dexmedetomidine
* Contraindication for moderate sedation in general

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of procedural sedation, using the 6 point Procedural Sedation State Scale PSSS | Initiation of procedure, around 30 minutes after medication was given
  Primary outcome is target sedation state measured with the PSSS (Pediatric Sedation State Scale) at initiation of the procedure, assessed via videotape by two independent research assistants. This scale has been developed and validated to reflect behaviours associated with adequate and inadequate sedation, in addition to adverse events associated with excessive sedation. States are predefined and related to the numbers 0 to 5. State 2 and 3 are defined as target sedation state. Primary outcome are number of patients in target sedation state.

SECONDARY OUTCOMES:
Anxiety relief, measured with a validated 18-points-observer score | Baseline, positioning for procedure, initiation of procedure, end of procedure
  mYPAS-SF (Modified Yale Preoperative Anxiety Scale Short Form) is a validated anxiety scale in pediatric sedation. Scores range from 4 to 18, with 18 being the highest level of anxiety. Lower scores are a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Hoeffe, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern

IPD SHARING:
Plan to Share IPD: No